CLINICAL TRIAL: NCT05358782
Title: The Influence of Implant Position on the Occurrence of Biological Complications: a Retrospective, Observational Study on Periapical Radiographs
Brief Title: The Influence of Implant Position on the Occurrence of Biological Complications
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: IMP-MAL
Record Dates: First submitted 2022-04-28; First posted 2022-05-03 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Peri-Implantitis
Keywords: peri-implant loss; dental radiography; implant malposition
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Implant with peri-implantitis: Implant with progressive marginal bone loss
  Interventions: Device: Dental implant positioning
- Healthy implant: Implant without any sign of marginal bone loss
  Interventions: Device: Dental implant positioning

INTERVENTIONS:
Device: Dental implant positioning — observational study of the effect of implant malposition

SUMMARY:
The primary objective of this study will be to study the correlation between implant position (malposition), evaluated through periapical radiographs of peri-implantitis vs healthy implants, and the occurrence of peri-implant biological complications such as peri-implantitis, as evaluated after at least 6 months from the placement of the prosthesis. The clinical records of all subjects treated with implants during the period between January 1st, 2005, and June 30th, 2021 (last follow-up included: 6 month visit on December 2021) in the Dental Clinic of the IRCCS Istituto Ortopedico Galeazzi (Milan, Italy) will be screened for inclusion.

Will be included 45 implants with peri-implantitis and 135 healthy implants regardless of the corresponding number of patients . Descriptive statistics will be provided by means of mean values and standard deviations. Correlation between baseline parameters and outcomes will be measured through regression analysis, being the independent variable the occurrence of peri-implantitis. Multilevel analysis will be performed.

For all the analysis, the level of significance was set at p<0.05.

For sample size calculation the investigators have considered alpha = .05, power = 80% and a proportion between controls and cases of 3:1. The investigators hypothesized a detection of an effect of malposition with a proportion of 0.25 of exposes in control group and 0.5 in test group. the investigators decided to include 45 implants with peri-implantitis and 135 healthy implants, after augmenting the numbers hypothesizing a maximum of 10% dropouts. The proportion of exposed are estimated on the basis of the study published by Yi et al. in 2020 .

The calculation was performed using the method proposed by Schoenfeld.

DETAILED DESCRIPTION:
The primary outcome was the occurrence of peri-implantitis described as:

* presence of signs of inflammation (bleeding and / or suppuration after probing);
* radiographic bone loss in addition to crestal bone resorption caused by initial remodeling or, in the absence of radiography at one year, bone level positioned ≥ 3 mm apically to the most coronal portion of the intraosseous portion of the implant body;
* presence of increased probing depth as compared to previous measurements, if available.

Implant malposition will be defined on the basis of the following parameters:

* criteria proposed by Buser and coworkers in 2004: at least 1.5 - 2 mm between implant neck and adjacent tooth (mesio-distal); ii) at least 1 mm of apico-coronal distance between implant neck and the Cemento-enamel Junction (CEJ) of adjacent teeth (no more than 2.5 mm); iii) at least 3 mm between the necks of two adjacent implants.
* inclination of the implant axis as compared the axis of adjacent teeth (both mesial and distal if present)
* characteristics of the prosthesis (emergency profile, presence of cantilevers, imprecise implant-abutment connection)

The following parameters will be collected from clinical records:

* implant-related factors: implant type, length, diameter, and type of implant-abutment connection, implant surface, vertical position of the implant (distance between implant neck and the bone level at the time of intervention (I-BC) (periapical radiograph)), distance between the implant neck margin and adjacent teeth (on periapical radiographs) (I-MT, I-DT [I-MI, I-DI]), distance between implant neck and the projection of CEJ of adjacent teeth (periapical radiographs) (I-MT-CEJ, I-DT-CEJ), the angle between the projection of the implant axis and the axis of adjacent teeth or implant.
* patient-related factors: age, gender, smoking status, systemic disease, medications, presence of periodontal disease at the time of intervention (severity), history of periodontal disease, bruxism;
* site-related factors: implant position / site, bone quantity / quality following the Lekholm and Zarb classification;
* prosthesis-related factors (to be evaluated using the radiographs taken after placement of the prosthesis): single crown, partial fixed denture, ceramic- or resin-made, time of loading, fixation methods (screwed or cemented), platform switching, crown height (I-CH), extension of prosthetic cantilever (only for single-tooth restorations) (mesial and / or distal) (C-M, C-D), angle of emergency profile (mesial and distal) (C-M-EP, C-D-EP), presence of misfit of the prosthesis.

Clinical data will be completely anonymized through the association of each subject to one identification code, and the elimination of the document containing the link between them.

ELIGIBILITY:
Inclusion Criteria:

* subjects aged more than 18 years old, treated with implants with moderately rough surface.
* subjects treated with dental implants at Istituto Ortopedico Galeazzi during the period between January 1st, 2005, and June 30th, 2021
* subjects without any systemic disease that could be an impact on bone metabolism (e.g. diabetes mellitus, osteoporosis, neoplasms)
* single and partial rehabilitations (without cantilever extension): single tooth restorations (one implant between two teeth or one single implant supporting single-tooth prosthesis with one adjacent tooth); multiple tooth restorations (one tooth per implant or bridges, splinted or not).
* complete information about patient status (systemic diseases, smoking status, medications, age, gender)
* complete description of the surgical and prosthetic protocol that was adopted.
* at least one periapical radiograph of good quality taken at the end of the intervention and a sufficient number of follow-up visits (at least one per year); the quality of the images will be assessed by the Guidance Notes for Dental Practitioners on the Safe Use of X-Ray Equipment ((UK) 2018), accepting Grade 1 and Grade 2 images.
* having clinical and / or radiographic records to assess periodontal status at the time of intervention.

Exclusion Criteria:

* Incomplete data (e.g. absence of periapical radiographs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The clinical records of all subjects treated with implants during the period between January 1st, 2005, and June 30th, 2021 (last follow-up included: 6 month visit on December 2021) in the Dental Clinic of the IRCCS Istituto Ortopedico Galeazzi (Milan, Italy) will be screened for inclusion.
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2022-04-06 (Actual); Primary Completion 2022-10-06 (Estimated); Study Completion 2023-02-06 (Estimated)

PRIMARY OUTCOMES:
occurence of peri-implantitis | 198 months
  Correlation between implant position (malposition), evaluated through periapical radiographs of peri-implantitis vs healthy implants, and the occurrence of peri-implant biological complications such as peri-implantitis

SECONDARY OUTCOMES:
occurence of peri-implantitis independently from smoking/periodontitis | 198 months
  assess how implant position is related to the occurrence of peri-implantitis, independently from the exposure to smoking or to periodontitis
operator's experience | 198 months
  the influence of operator's experience on the odds of development of peri-implantitis
implant-tooth and implant-implant distance | 198 months
  - the occurrence of peri-implantitis as related to absolute values of implant-tooth and implant-implant distance
characteristics of the prosthesis | 198 months
  - the occurrence of peri-implantitis as related to characteristics of the prosthesis (emergency profile, cantilevers, imprecise implant-abutment connection)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Quality assessment of radiographs. 2018. London: FGDP(UK); [accessed]. https://www.fgdp.org.uk/SiD/a2-quality-assessment-radiographs.
- [Background] Arunyanak SP, Sophon N, Tangsathian T, Supanimitkul K, Suwanwichit T, Kungsadalpipob K. The effect of factors related to periodontal status toward peri-implantitis. Clin Oral Implants Res. 2019 Aug;30(8):791-799. doi: 10.1111/clr.13461. Epub 2019 Jun 12. PMID 31107993
- [Background] Berglundh T, Armitage G, Araujo MG, Avila-Ortiz G, Blanco J, Camargo PM, Chen S, Cochran D, Derks J, Figuero E, Hammerle CHF, Heitz-Mayfield LJA, Huynh-Ba G, Iacono V, Koo KT, Lambert F, McCauley L, Quirynen M, Renvert S, Salvi GE, Schwarz F, Tarnow D, Tomasi C, Wang HL, Zitzmann N. Peri-implant diseases and conditions: Consensus report of workgroup 4 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Clin Periodontol. 2018 Jun;45 Suppl 20:S286-S291. doi: 10.1111/jcpe.12957. PMID 29926491
- [Background] Buser D, Martin W, Belser UC. Optimizing esthetics for implant restorations in the anterior maxilla: anatomic and surgical considerations. Int J Oral Maxillofac Implants. 2004;19 Suppl:43-61. PMID 15635945
- [Background] Canullo L, Tallarico M, Radovanovic S, Delibasic B, Covani U, Rakic M. Distinguishing predictive profiles for patient-based risk assessment and diagnostics of plaque induced, surgically and prosthetically triggered peri-implantitis. Clin Oral Implants Res. 2016 Oct;27(10):1243-1250. doi: 10.1111/clr.12738. Epub 2015 Nov 20. PMID 26584716
- [Background] Ferreira SD, Martins CC, Amaral SA, Vieira TR, Albuquerque BN, Cota LOM, Esteves Lima RP, Costa FO. Periodontitis as a risk factor for peri-implantitis: Systematic review and meta-analysis of observational studies. J Dent. 2018 Dec;79:1-10. doi: 10.1016/j.jdent.2018.09.010. Epub 2018 Nov 2. PMID 30391683
- [Background] Francetti L, Cavalli N, Taschieri S, Corbella S. Ten years follow-up retrospective study on implant survival rates and prevalence of peri-implantitis in implant-supported full-arch rehabilitations. Clin Oral Implants Res. 2019 Mar;30(3):252-260. doi: 10.1111/clr.13411. Epub 2019 Feb 18. PMID 30702771
- [Background] Lekholm U, Zarb GA. 1985. Patient selection and preparation. In: Branemark PI, Zarb GA, Albrektsson T, editors. Tissue-integrated prostheses: Osseointegration in clinical dentistry. Chicago: Quintessence. p. 199-209.
- [Background] Monje A, Aranda L, Diaz KT, Alarcon MA, Bagramian RA, Wang HL, Catena A. Impact of Maintenance Therapy for the Prevention of Peri-implant Diseases: A Systematic Review and Meta-analysis. J Dent Res. 2016 Apr;95(4):372-9. doi: 10.1177/0022034515622432. Epub 2015 Dec 23. PMID 26701350
- [Background] Schoenfeld DA. Sample-size formula for the proportional-hazards regression model. Biometrics. 1983 Jun;39(2):499-503. PMID 6354290
- [Background] Yi Y, Koo KT, Schwarz F, Ben Amara H, Heo SJ. Association of prosthetic features and peri-implantitis: A cross-sectional study. J Clin Periodontol. 2020 Mar;47(3):392-403. doi: 10.1111/jcpe.13251. Epub 2020 Jan 21. PMID 31912511